CLINICAL TRIAL: NCT03877497
Title: To Reach Unrestricted Services for Transgender Women
Acronym: TRUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Florida International University (Other)
Responsible Party: Principal Investigator, Elena Cyrus, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K99/R00 DA046311
Record Dates: First submitted 2018-12-06; First posted 2019-03-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Transgender Women; Substance Abuse; Hiv
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SBIRT-T (Experimental): The screening, brief intervention and referral to treatment (SBIRT-T) will be adapted and used as the intervention in the experimental arm
  Interventions: Behavioral: Adapted SBIRT-T for transgender women
- INFO-C (Active Comparator): The INFO-C group is a time-matched comparison control where information will be provided on substance use and PrEP services in a non-SBIRT-T format via printed and audio-visual study material
  Interventions: Behavioral: Adapted SBIRT-T for transgender women

INTERVENTIONS:
Behavioral: Adapted SBIRT-T for transgender women — Transgender women will be screened for substance use. Those at moderate risk or less will be randomized into the study into either the intervention arm (SBIRT-A) or the control arm (CONTROL-C). Those at higher risk will be ineligible for the study and referred for substance use treatment services
  Other Names: SBIRT-T

SUMMARY:
Florida has the fifth largest transgender population in the United States. Transgender women, particularly those of color, in the southern part of Florida are a marginalized population who are impacted by co-morbidities of substance abuse and HIV in their communities. The overall objective of the study is to use a vetted adapted brief intervention to stem the development of substance abuse in at-risk transgender women, and thereby increase primary and secondary prevention methods such as routine HIV screening, uptake of pre-exposure prophylaxis (PrEP) and use of non-occupational post-exposure prophylaxis (nPEP).

DETAILED DESCRIPTION:
Background: Transgender women are disproportionally affected by substance abuse and HIV. Evidence-based interventions that can address both issues simultaneously may efficiently improve the overall health of transgender women and reduce burdensome health and societal costs associated with substance abuse and HIV. In South Florida, the majority of transgender women identify as Black or Latina, or transgender women of color (TWOC). TWOC are at highest risk for substance abuse and HIV acquisition, due to multiple external stressors arising as a consequence of being a gender minority, and also a racial/ethnic minority. Studies have demonstrated Screening, Brief Intervention, and Referral to Treatment (SBIRT) to be effective in mitigating development of substance use disorders (SUD) in other at-risk, marginalized populations. An adapted culturally-tailored SBIRT focused on linkage to substance use services and HIV pre- and post-exposure prophylaxis (PrEP and nPEP) may effectively reduce the odds of individuals in this special population developing a SUD and also facilitate their voluntary election of HIV screening and use of PrEP/nPEP for HIV prevention. Objectives: K99 -In preparation for the independent phase, the career development phase will include training in qualitative research methods and intervention development. R00 - In the independent phase, the study objectives will be to (a) use a mixed-methods approach to obtain formative data among 40 transgender women that will aid in adapting and developing an adapted culturally tailored SBIRT intervention (SBIRT-A), (b) pre-test and refine SBIRT-A in 15 transgender women based on formative work and, (c) pilot test SBIRT-A in a sample of 76 transgender to assess feasibility and acceptability. Pilot Design: Randomized trial among 76 adult (18 years or older) HIV uninfected transgender women at moderate risk for developing a substance use disorder who will be randomized to either SBIRT-A or the control condition (INFO-C). The INFO-C group will be a time-matched comparison control where information will be provided on substance use and PrEP services in a non-SBIRT format via printed and audio-visual study material. There will be a follow-up visit in three months to assess linkage, and barriers and facilitators to substance use services and PrEP/nPEP. Analysis: Bivariate difference tests (chi square and t-tests) will be used to test differences between SBIRT-A and INFO-C participants for the primary outcome measures (linkage to substance use services, PrEP, and nPEP) at the three-month visit. Multivariate binary logistic regressions (post- and pre-intervention) will be used to determine substance use as a predictor of (1) HIV/STI screening in the past three months and (2&3) PrEP and nPEP uptake in the past three months. Significance: Results derived from this study will help elucidate the relationship between substance use and HIV among transgender women, including TWOC, in South Florida, and will provide evidence for a larger study that can test the efficacy of SBIRT-A to reduce prevalence of substance abuse and HIV in this special population. The aims of this study are parallel to the NIH/National Institute on Drug Abuse (NIDA) strategic plan to decrease HIV/AIDS health disparities, prevent HIV transmission, and better understand the interaction of drug abuse and HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Transgender woman over the age of 18
* HIV uninfected
* no current substance abuse use according to AUDIT and SBIRT criteria

Exclusion Criteria:

* HIV infected transgender woman
* evidence of hazardous alcohol or illicit drug use

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women
Enrollment: 86 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with substance abuse | 6 months
  The rate of change of substance abuse incidence for both arms

SECONDARY OUTCOMES:
Rate of Preexposure prophylaxis (PrEP) election | 6 months
  The rate of PrEP election (or new PrEP users) among study participants in both arms

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida International University, Miami, Florida
  - University of Central Florida, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided